CLINICAL TRIAL: NCT05385562
Title: Formulated Posterior Subtenon Triamcinolone (PSTA) Injection Versus Posterior Subtenon Triamcinolone Alone in the Management of Macular Edema Secondary to Non-ischemic Retinal Vein Occlusions
Brief Title: Formulated PSTA Injection Versus PATA Alone in the Management of Macular Edema Secondary to Non-ischemic Retinal Vein Occlusions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Ehab tharwat, Dr, Al-Azhar University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PSTA and macular edema
Record Dates: First submitted 2022-05-18; First posted 2022-05-23 (Actual); Last update posted 2022-05-26 (Actual); Status verified 2022-05

CONDITIONS: Macula Edema
MeSH Terms: interventions — Triamcinolone Acetonide; Hyaluronic Acid; Chondroitin Sulfates

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Formulated Posterior Sub Tenon Triamcinolone (Active Comparator)
  Interventions: Drug: Triamcinolone Acetonide and sodium hyaluronate and chondroitin sulfate
- Posterior Sub Tenon Triamcinolone alone (Active Comparator)
  Interventions: Drug: Triamcinolone Acetonide alone

INTERVENTIONS:
Drug: Triamcinolone Acetonide and sodium hyaluronate and chondroitin sulfate — formulated with sodium hyaluronate and chondroitin sulfate
  Arms: Formulated Posterior Sub Tenon Triamcinolone
Drug: Triamcinolone Acetonide alone — Triamcinolone Acetonide alone
  Arms: Posterior Sub Tenon Triamcinolone alone

SUMMARY:
The aim of this study is to compare formulated Posterior Subtenon Triamcinolone acetonide (PSTA) injection versus Posterior Subtenon Triamcinolone acetonide alone in the management of macular edema secondary to non-ischemic retinal vein occlusions, either central or branch.

ELIGIBILITY:
Inclusion Criteria:

* Diminution vision due to macular edema secondary to non-ischemic retinal vein occlusions, either central or branch, as evidenced by clinical and angiographic evaluation
* CMT ≥ 250 µ.
* Willing to participate in the study

Exclusion Criteria:

* Unwilling to participate in the study.
* Ischemic RVO
* Prior laser treatment
* Glaucoma/Ocular Hypertension
* Cataract which lead to difficulty in the evaluation of macula
* Vitreous hemorrhage
* Macular ischemia
* Iris neovascularisation
* patients with intravitreal injection of anti VEGFs, steroid, or any intraocular surgery 3 months prior to the inclusion.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2020-01-02 (Actual); Primary Completion 2022-05-01 (Actual); Study Completion 2022-05-10 (Actual)

PRIMARY OUTCOMES:
Best-corrected visual acuity (BCVA) | Baseline
  will be measured with the Snellen chart
Best-corrected visual acuity (BCVA) | at 1st month
  will be measured with the Snellen chart
Best-corrected visual acuity (BCVA) | at 3rd month
  will be measured with the Snellen chart
Best-corrected visual acuity (BCVA) | at 6th month
  will be measured with the Snellen chart
central macular thickness ( CMT) | at baseline
  CMT will be measured with OCT
central macular thickness ( CMT) | at 1st month
  CMT will be measured with OCT
central macular thickness ( CMT) | at 3rd month
  CMT will be measured with OCT
central macular thickness ( CMT) | at 6th month
  CMT will be measured with OCT

CONTACTS AND LOCATIONS:
Locations (1):
- Ehab tharwat, Damietta, New Damietta, Egypt

IPD SHARING:
Plan to Share IPD: Undecided